CLINICAL TRIAL: NCT05559814
Title: Intraluminal Peppermint Oil Can Increase Adenoma Detection Rate in Colon Cancer Screening Colonoscopy: A Double- Blinded Randomized Controlled Trial
Brief Title: Intraluminal Peppermint Oil and Adenoma Detection Rate in Screening Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: The Royal College of Physicians of Thailand (Unknown)
Responsible Party: Principal Investigator, Uayporn Kaosombatwattana, Department of Medicine, Siriraj Hospital, Mahidol university, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: Si 098/2021
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Colonic Polyp
Keywords: Peppermint oil, Adenoma detection rate, Colonic peristalsis
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peppermint oil (Experimental): 1.6% peppermint oil solution 50 ml(Peppermint oil plus simethicone and tween)
  Interventions: Drug: Intraluminal peppermint oil
- Placebo (Placebo Comparator): Placebo solution 50ml(Simethicone plus tween)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intraluminal peppermint oil — Intraluminal flushing of peppermint oil solution through the scope channel during the scope withdrawal
  Arms: Peppermint oil
Drug: Placebo — Intraluminal flushing of placebo solution through the scope during scope withdrawal
  Arms: Placebo

SUMMARY:
This is a prospective randomized placebo-controlled trial to evaluate the efficacy of peppermint oil spraying into the colonic lumen through the scope channel during screening colonoscopy. The primary outcome is to compare the colonic peristalsis between peppermint oil and placebo. The secondary outcomes compare the procedural time, polyp detection rate, adenoma detection rate, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

- Participants with age > 18 years who attended for colorectal cancer screening colonoscopy.

Exclusion Criteria:

* Participants who had been colectomy
* Participants who diagnosed of inflammatory bowel disease or polyposis syndrome.
* Participants who had been took anti-spasmosic drugs prior to colonoscopy within 24 hours (Anticholibergic/Antimuscarinic : Hyoscine(Buscopan®), Dicyclomine(Berclomine®) or Smooth muscle relaxant : Mebeverine(Duspatin®,Colofac®), Pinaverium bromide(Dicetel®), Alverine(Meteospasmyl®), Peppermint oil(Colpermin®))
* Participants with Prothrombin time > 3 second ULN, INR > 1.5 or Platelet < 50,000.
* Pregnancy or breast feeding
* Participants who cannot consent.
* Participants who had history of peppermint oil allergy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate(ADR) | During colonoscopy
  Number of adenoma per total participants who were colonoscopy in both groups

SECONDARY OUTCOMES:
Adenoma per posititive participants(APP) | During colonoscopy
  Number of aenama in patients who had found at least one adenoma in both groups
Colonic peristalsis grading | During colonoscopy
  Percentage of colonic peristalsis grade 0 and 1 in peppermint oil group in both groups
Time of polyps resection | During colonoscopy
  Time of polypectomy per polyp in both groups
Intravenous anti-spasmodic agents | During colonoscopy
  Percentage of intravenous anti-spasmodic agents in both groups
Adeverse events | 24 hours after colonoscopy
  Total number of adverse events in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of internal medicine siriraj hospital, Mahidol university, Bangkok Noi, Bangkok, Thailand